CLINICAL TRIAL: NCT06389474
Title: A Phase III Study to Evaluate the Efficacy of INM004 (Shiga Antitoxin) in Pediatric Patients With Shiga Toxin-producing Escherichia Coli-associated Hemolytic Uremic Syndrome.
Brief Title: Efficacy of INM004 in Children With STEC-HUS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Inmunova S.A. (Other)
Collaborators: Exeltis (Industry); Chemo Research (Industry); Linical (Unknown); KLIXAR (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-INM004-04
Record Dates: First submitted 2024-04-25; First posted 2024-04-29 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Hemolytic-Uremic Syndrome
Keywords: STEC-HUS; Typical Hemolytic Uremic Syndrome; Diarrhea asociated-Hemolytic Uremic Syndrome; Shiga toxin-producing Escherichia coli; Shiga toxin
MeSH Terms: conditions — Hemolytic-Uremic Syndrome | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Adaptive design. IA will be done when approximately 50% of the enrollment is reached and the participants have completed 28 days of follow-up. This analysis will not be blinded and will be carried out to declare futility or re-estimate the sample size. The re-estimation of the sample size will allow a maximum of 300 randomized subjects in total, but a reduction in the initial item size of 220 subjects is not expected. In case of re-estimating the sample size, the smallest sample size under 300 will be selected, which allows a power of ≥ 80%. %. If with 300 subjects, a power of 80% is not reached, but it is ≥ 50%, then the sample size is re-estimated to 300 subjects, as long as the conditional power of the IA is ≥ 50% (promising results)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- INM004 (Experimental): Two doses of Anti-Shiga Toxin Hyperimmune Equine Immunoglobulin F(ab´)2 fragment at a dosage of 4 mg/kg of body weight, 24 hours apart.
  Interventions: Biological: INM004
- Placebo (Placebo Comparator): Two doses of saline solution, 24 hours apart.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: INM004 — Two doses of Anti-Shiga Toxin Hyperimmune Equine Immunoglobulin F(ab´)2 fragments at a dosage of 4 mg/kg of body weight, 24 hours apart. Each vial contains 25 mg of protein/ml. Therefore, each subject must receive 0.16 ml/kg per dose. The vial volume will be reconstituted in a 100 ml (for subjects with a body weight of 20 kg or more) or 50 ml (for subjects under 20 kg of body weight) infusion bag. It will be administered as an intravenous infusion using an infusion pump over a period of 50 minutes. In subjects with a BMI over 30 kg/m2, infusion will be performed over a period of 100 minutes
  Other Names: Active
  Arms: INM004
Other: Placebo — Two doses of placebo, 24 hours apart. The placebo solution has the same composition of excipients as INM004 without the active pharmaceutical ingredient, and its appearance is identical. Each subject must receive 0.16 ml/kg of placebo solution per dose. The vial volume will be reconstituted in a 100 ml (for subjects with a body weight of 20 kg or more) or 50 ml (for subjects under 20 kg of body weight) infusion bag. It will be administered as an intravenous infusion using an infusion pump over a period of 50 minutes. In subjects with a BMI over 30 kg/m2, infusion will be performed over a period of 100 minutes
  Other Names: Control
  Arms: Placebo

SUMMARY:
The objectives of this study are to evaluate the efficacy, safety, and pharmacokinetics of INM004 in pediatric patients with Hemolytic Uremic Syndrome associated to infection by Shiga toxin-producing Escherichia coli (STEC-HUS).

DETAILED DESCRIPTION:
The primary objective will be to evaluate the efficacy of INM004, added to the standard of care, as a treatment for STEC-HUS in the amelioration of renal function.

Secondary objectives

* To evaluate the efficacy of INM004 in the reduction of mortality.
* To evaluate the efficacy of INM004 in the prevention and reduction of extrarenal complications.
* To evaluate the efficacy of INM004 in the improvement of TMA laboratory parameters.
* To evaluate the efficacy of INM004 in the reduction of hospital stay days.
* To evaluate the safety of INM004
* To evaluate the pharmacokinetics of INM004
* To evaluate the kinetics of Stx

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 9 months and < 18 years at the time of randomization.
2. In addition, only for subjects < 1 year and ≥ 15 years, confirmation of STEC infection determined by:

   1. Detection of generic Stx, Stx1, Stx2, or Stx1/Stx2 in stools by enzyme immunoassay (EIA); or
   2. Detection of stx, stx1, stx2, or stx1/stx2 genes in stools by Polymerase Chain Reaction (PCR); or
   3. Detection of specific anti-polysaccharide (IgM) antibodies in serum; or
   4. Fecal culture positive for E. coli O157 confirmed by serogroup-specific seroagglutination.
3. Hospitalization at the participating institution.
4. History of onset of diarrhea within 10 days prior to STEC-HUS diagnosis at the participating institution.
5. Diagnosis of STEC-HUS defined as a subject with signs of renal damage, hemolysis, and platelet consumption:

   1. Signs of renal damage defined as:

      * Serum creatinine value above the ULN for age and sex, and GFR below the LLN for age, sex, and height.
   2. Presence of hemolysis documented by:

      * LDH levels above the ULN for age, and/or
      * Presence of schistocytes in peripheral blood smear.
   3. Platelet consumption according to any of the following laboratory criteria:

      * Peripheral blood platelet count < 150 × 103/μL, and/or
      * A ≥50% decrease in peripheral blood platelet count compared to a sample collected within the previous 24 hours.
6. Informed consent form signed and dated by the subject or, the legal guardian(s), with the subject's assent as appropriate based on age and regulatory guidelines in the region.
7. Subjects who have already had menarche must have a negative pregnancy test.

Exclusion Criteria:

1. Start of dialysis within 48 hours prior to admission to the participating institution.
2. More than 24 hours from diagnosis of STEC-HUS at the participating institution up to randomization.
3. History of chronic/recurrent hemolytic anemia, thrombocytopenia, or CKD.
4. Personal and/or family history of atypical HUS.
5. Suspected HUS secondary to infectious processes other than gastrointestinal (e.g., Streptococcus pneumoniae, HIV).
6. Suspected HUS secondary to other etiologies (e.g., drug-associated HUS, neoplasms, bone marrow or solid organ transplantation, autoimmune disorders).
7. Any other acute or chronic medical condition that, in the opinion of the investigator, may interfere with the evaluation of the efficacy and/or safety of the study medication.
8. History of: a) anaphylaxis of any kind; b) prior administration of equine serum (e.g., antivenom, anti-arachnid serum, anti-SARS-CoV-2 serum, etc.) or an allergic reaction from contact or exposure to horses.
9. Pregnant or breastfeeding woman.
10. Impossibility of hospitalization in the participating institution.
11. Concurrent participation in another clinical trial or having participated in a clinical trial in the last 3 months.
12. Severe malnutrition. Defined when the weight is three standard deviations below the median, according to height, age and sex as per WHO guidelines.
13. Medical conditions that may affect kidney function or cause/enhance neurological symptoms or signs:

    * Congenital or acquired anomalies that may affect functioning renal mass.
    * Epilepsy or structural abnormalities of the brain that may increase the risk of seizures.
    * Trisomy 21.
    * Prematurity (born before 28 weeks gestation).
    * Other (according to investigator criteria).

Ages: 9 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 220 (Estimated)
Dates: Start 2024-10-05 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to recovery of renal function during the acute phase | 28 days
  Time (days) to achieve a glomerular filtration rate greater than or equal to the lower limit of normal (according to age, height, and sex) and a serum creatinine lower than or equal to the upper limit of normal (according to age and sex), both measured in the absence of dialysis.

SECONDARY OUTCOMES:
Short-term recovery of renal function | 90 days
  Proportion of subjects with a glomerular filtration rate ≥ lower limit of normal (according to age, height and sex) and serum creatinine ≤ upper limit of normal (according to age and sex), both measured in the absence of dialysis.
MAKE 90 | 90 days
  Proportion of subjects meeting any of the following criteria at day 90: death, dialysis requirement after 24 hours post-randomization, dialysis of more than 10 days, or persistent decline in renal function (without recovery of glomerular filtration rate according to age, height, and sex).
Dialysis longer than 10 days | 90 days
  Proportion of dialyzed subjects requiring more than 10 days of dialysis
Dialysis requirement | 90 days
  Proportion of subjects requiring dialysis after 24 hours post-randomization
Mortality | 90 days
  Proportion of subjects who die from any cause.

OTHER OUTCOMES:
CKD Risk Assessment According to Kidney Disease Improving Global Outcomes (KDIGO) Categories | 90 days
  Proportion of subjects in each CKD category (low, medium, high, very high) according to GFR and albuminuria at day 90
Evolution of renal function at 7 days (GFR_AUC1-7) | 7 days
  Area under the curve of glomerular filtration rate from Day 1 to Day 7
Evolution of renal function at 28 days (GFR_AUC1-28) | 28 days
  Area under the curve of glomerular filtration rate from Day 1 to Day 28
Evolution of renal function at 90 days (GFR_AUC1-90) | 90 days
  Area under the curve of glomerular filtration rate from Day 1 to Day 90
Incidence of anuria | 90 days
  Proportion of subjects with anuria onset after 24 hours post-randomization
Extrarenal composite endpoint | 90 days
  Proportion of subjects who develop at least one severe extrarenal event including neurological events (coma, seizure, stroke), cardiovascular (hemodynamic instability, heart failure, acute myocardial infarction, myocarditis), respiratory (respiratory distress), gastrointestinal (hemorrhagic colitis, intestinal necrosis, intussusception, pancreatitis, severe hepatitis) or death.
Recovery of the thrombotic microangiopathy (TMA), thrombocytopenia | 90 days
  Normalization of thrombocytopenia (platelet count ≥150,000/mm3), measured as time to recovery.
Recovery of the thrombotic microangiopathy (TMA), hemolytic anemia | 90 days
  Proportion of subjects with recovery from hemolytic anemia (Hemoglobin ≥ lower limit of normal and Lactate Dehydrogenase ≤ upper limit of normal).
Duration of hospitalization | 90 days
  Time from randomization to hospital discharge.
Incidence of adverse events of special interest | 28 days
  * Incidence of injection site reactions.
  * Incidence of hypersensitivity (i.e., allergic reaction, anaphylaxis and serum sickness)
Incidence of adverse events | 90 days
  Incidence of adverse events
Pharmacokinetic - AUC0-t | 144 hours
  Area under the curve of INM004 concentration from time 0 to the last measurable concentration
Pharmacokinetic - AUC0-inf | 144 hours
  Area under the curve of INM004 concentration as a function of time extrapolated to infinity
Pharmacokinetic - Cmax | 144 hours
  Maximum concentration of INM004 in plasma after administration
Pharmacokinetic - Tmax | 144 hours
  Time in which INM004 reaches the maximum concentration in plasma after administration
Pharmacokinetic - λz | 144 hours
  Terminal velocity constant via linear logit regression
Pharmacokinetic - t1/2 | 144 hours
  Terminal half-life of INM004
Pharmacokinetic - Vz | 144 hours
  Volume of distribution of INM004
Pharmacokinetic - Cl | 144 hours
  INM004 clearence
Pharmacokinetic - AUC/dose | 144 hours
  Area under the curve of INM004 normalized for the administered dose
Pharmacokinetic - Cmax/dose | 144 hours
  Maximum concentration of INM004 in plasma normalized for the administered dose
Baseline Shiga toxin serum levels | Baseline
  Baseline serum Stx2 concentration in all subjects
Kinetics of Shiga toxin in serum | 144 hours
  Serum Stx2 concentration at different time-points in placebo subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Sanguineti, Ph.D, Study Director — Inmunova S.A.
Locations (52):
- Argentina (25):
  - Hospital Interzonal Dr. José Penna, Bahía Blanca, Buenos Aires
  - Hospital Penna, Bahía Blanca, Buenos Aires
  - Hospital de niños Sor María Ludovica, La Plata, Buenos Aires
  - Clinica del niño y la madre, Mar del Plata, Buenos Aires
  - Hospital Interzonal Especializado Materno Infantil Don Victorio Tetamanti, Mar del Plata, Buenos Aires
  - Sanatorio de la Trinidad Ramos Mejia, Ramos Mejía, Buenos Aires
  - Hospital El Cruce, San Juan Bautista, Buenos Aires
  - Sanatorio Güemes, Buenos Aires, Buenos Aires F.D.
  - Hospital de Pediatría S.A.M.I.C. "Prof. Dr. Juan P. Garrahan", Buenos Aires, Buenos Aires F.D.
  - Hospital General de Niños Pedro de Elizalde, Buenos Aires, Buenos Aires F.D.
  - Sanatorio Anchorena, CABA, Buenos Aires F.D.
  - Hospital Privado Centro Médico de Córdoba, Córdoba, Córdoba Province
  - Hospital de Niños de la Santísima Trinidad, Córdoba, Córdoba Province
  - Hospital "San Antonio de Padua" Río Cuarto, Río Cuarto, Córdoba Province
  - Hospital Pediátrico Dr. Humberto Notti, Mendoza, Mendoza Province
  - Hospital Teodoro J. Schestakow, San Rafael, Mendoza Province
  - Clínica Pediátrica San Lucas, Neuquén, Neuquén Province
  - Hospital Público Materno Infantil, Salta, Salta Province
  - Hospital Pediátrico San Luis, San Luis, San Luis Province
  - Hospital de Niños Zona Norte "Dr. Roberto M. Carra", Rosario, Santa Fe Province
  - Sanatorio de Niños, Rosario, Santa Fe Province
  - Hospital De Clínicas Pte. Nicolás Avellaneda, San Miguel de Tucumán, Tucumán Province
  - Clínica Zabala, Ciudad Autonoma de Buenos Aire
  - Hospital de Niños Dr. Ricardo Gutierrez, Ciudad Autonoma de Buenos Aire
  - Sanatorio Allende, Córdoba
- Cliniques universitaires Saint-Luc, Brussels, Belgium
- France (8):
  - CHU De Bordeaux, Bordeaux
  - Hospices Civils De Lyon - Hopital Femme Mere Enfant, Lyon
  - Centre Hospitalier Universitaire De Montpellier, Montpellier
  - CHU Nantes, Nantes
  - Hospital Necker Enfants Malades, Paris
  - Robert Debre University Hospital, Paris
  - Trousseau Hospital, Paris
  - CHU Rouen, Rouen
- Germany (3):
  - Charité - Universitätsmedizin Berlin, Berlin
  - University Hospital Cologne AöR, Cologne
  - Universitaetsklinikum Heidelberg AöR, Heidelberg
- Children's Health Ireland, Dublin, Ireland
- Italy (5):
  - University Hospital Consorziale Policlinico, Bari
  - IRCCS Sant'Orsola, Bologna
  - Istituto Gianina Gaslini, Genova
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedale Università, Padua
- Romania (3):
  - Spitalul Clinic de Urgenta pentru Copii Marie Sklodowska Curie, Bucharest
  - Spitalul Clinic De Urgenta Pentru Copii Cluj-Napoca, Cluj-Napoca
  - Spitalul Clinic de Urgenta pentru Copii Louis Turcanu, Timișoara
- Spain (3):
  - Hospital Universitario De Cruces, Barakaldo
  - Hospital Infantil Universitario Niño Jesus, Madrid
  - Hospital Universitario 12 De Octubre, Madrid
- United Kingdom (3):
  - Bristol Royal Hospital for Children, Bristol
  - Royal Hospital for Sick Children, Glasgow
  - Great Ormon Street Hospital for Children, London